CLINICAL TRIAL: NCT04014231
Title: A Novel Single Wave Assessment to Measure Cardiac Dysfunction and Metabolic Syndrome in Cancer Patients
Brief Title: Novel Single Wave Assessment in Measuring Cardiac Dysfunction and Metabolic Syndrome in Patients With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15317; NCI-2015-01612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15317 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2015-09-30; First posted 2019-07-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (single wave assessment): Patients undergo placement of a single wave application near the carotid region of the neck.
  Interventions: Procedure: Diagnostic Imaging; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Diagnostic Imaging — Undergo placement of single wave application
  Other Names: Medical Imaging
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies a novel single wave assessment in measuring cardiac dysfunction and metabolic syndrome in patients with cancer. The novel single wave assessment is a hand held device that can report left ventricular ejection fraction, which measures how well the heart is pumping blood (by giving a percentage) and measures how stiff the arteries are in the heart (pulse wave velocity). A novel single wave assessment may help identify patients at increased risk for type II diabetes and metabolic syndrome (disease where patients have increased blood pressure and high blood sugar level and excess body fat around the waist and abnormal cholesterol levels).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relationship between insulin resistance (delta omega) as measured by the single wave application and inflammation markers associated with insulin resistance and metabolic syndrome (MetS) in cancer patients, and to estimate the mean and standard deviation (sd) of delta omega in cancer patients with and without MetS for designing future, larger studies.

II. To determine the degree of agreement between the single wave measure of left ventricular ejection fraction (LVEF) in cancer patients and that measured by the routine 2-dimensional (2D) echocardiography (standard of care).

OUTLINE:

Patients undergo placement of a single wave application near the carotid region of the neck.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing 2D echocardiogram at City of Hope (COH)
* Patients with a current or past diagnosis of cancer
* Ability to sign a written informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Patients who have known "carotid sinus hypersensitivity"
* Patients who do not consent to blood draw
* Patients who have not fasted for the instructed time prior to blood draw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing 2D echocardiogram at City of Hope
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Single wave measure of insulin resistance (delta omega) and markers of inflammation | Up to end of single wave assessment
  The agreement of the single wave-based ejection fraction (EF) to EF measured by 2-dimensional (2D) echocardiography will be estimated in this study. Generalized linear models will be fitted to insulin resistance as the dependent variable and the inflammation markers as independent variables, adjusted for sex, age, and other clinical factors, along with an indicator of MetS (1 if present; 0 if absent) and the interactions of MetS and the inflammation markers to examine their association with insulin resistance.
Difference in left ventricular ejection fraction (LVEF) measured by the single wave application and 2D echocardiography | Up to end of single wave assessment
  Initially, the measurements from the two methods will be plotted to visualize their agreement. The Bland-Altman plot will then be used to assess the degree of agreement. The difference in LVEF measured by the two methods will be plotted against the mean of the measurements from the two methods. The 95% confidence interval for the mean difference will be determined. Sensitivity and specificity of the single wave-based LVEF measure for various cutpoints of LVEF from 2D echocardiography (as the gold standard) will also be computed. Pearson correlation coefficient will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne E Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States